CLINICAL TRIAL: NCT02197247
Title: A Phase I, Open-Label, Non-Randomised, Multicentre Study to Assess the Effect of Rifampicin (a CYP3A4 Inducer) on the Pharmacokinetics of AZD9291 in Patients With EGFRm Positive NSCLC Whose Disease Has Progressed on an EGFR TKI
Brief Title: Study to Assess the Effect of Rifampicin on Blood Levels and Safety of AZD9291, in Patients With EGFRm+ NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Other
Other Study IDs: D5160C00013; 2014-001525-32 (EudraCT Number)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: oncology, cancer, non small cell lung cancer, anticancer drug, pharmacokinetics, AZD9291, rifampicin, CYP P450 inducer, EGFR genes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifampicin and AZD9291 (Experimental): Sequential treatments of AZD9291 alone followed by AZD9291 +rifampicin, followed by AZD9291 alone.
  Interventions: Procedure: Pharmacokinetic sampling - AZD9291; Drug: Rifampicin; Drug: AZD9291 tablet dosing; Procedure: Pharmacokinetic sampling - rifampicin; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550

INTERVENTIONS:
Procedure: Pharmacokinetic sampling - AZD9291 — Blood sampling to measure AZD9291
Drug: Rifampicin — Rifampicin (CYP inducer) 600mg taken once daily from Day 29 to Day 49 (Part A)
Drug: AZD9291 tablet dosing — Part A: AZD9291 80mg tablet taken daily from Days 1 to 77. Part B: AZD9291 80mg tablet taken daily for 12 months.
Procedure: Pharmacokinetic sampling - rifampicin — Blood sampling to measure rifampicin levels
Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550 — Blood samples to measure levels of AZ5140 and AZ7550

SUMMARY:
This is a Phase I, open-label, 2-part study in patients with a confirmed diagnosis of epidermal growth factor receptor (EGFR) mutation positive (EGFRm+) non-small cell lung cancer (NSCLC), who have progressed following prior therapy with an approved EGFR tyrosine kinase inhibitor (TKI) agent.

Part A will assess the effect of rifampicin on the pharmacokinetic (PK) parameters of AZD9291 and metabolites AZ5104 and AZ7550 following multiple oral dosing of both rifampicin and AZD9291 in a fasted state.

Part B will allow patients further access to AZD9291 after the PK phase (Part A) and will provide for additional safety data collection. All patients who complete Part A will be able to enter part B, and continue to receive AZD9291 80 mg once daily until: disease progression; they are no longer deriving clinical benefit; or any other reason.

ELIGIBILITY:
For inclusion in the study patient should fulfil the following criteria:

1. Male or female, aged at least 18 years. 2. Histological or cytological confirmation diagnosis of NSCLC. 3. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI, eg gefitinib, erlotinib or afatinib. In addition, other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.

4. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).

5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks (Appendix G).

6. Patients must have a life expectancy of ≥12 weeks as estimated at the time of screening.

7. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments. Women under 50 years old would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.

8. Male patients should be willing to use barrier contraception, ie, condoms, until 6 months after last study drug is taken.

9. Contact lens wearers must be prepared to not wear contact lenses and wear glasses for the duration of the rifampicin dosing.

1. Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
2. Treatment with any of the following: Treatment with an EGFR TKI (eg, erlotinib or gefitinib) w/in 8 days or approx. 5 x half-life, whichever is the longer, of the first dose of study treatment; any cytotoxic chemo, investigational agents or other anticancer drugs from a previous treatment regimen w/in 14 days of the first dose of study treatment; major surgery (excluding placement of vascular access) w/in 4 weeks of the first dose of study treatment; radiotherapy with a limited field of radiation for palliation w/in 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of bone marrow or with a wide field of radiation which must be completed w/in 4 weeks of the first; patients currently receiving (or unable to stop use prior to receiving the first dose) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior). All patients must avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
3. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the final PK sample collection on Day 78 of Part A.
5. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and HIV. Screening for chronic conditions is not required.
7. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: ANC <1.5 x 10^9/L; Platelet count <100 x 10^9/L; Haemoglobin <90 g/L; ALT >2.5 times the ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; AST >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases; creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
8. Any of the following cardiac criteria: Mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor (QTcF) >470 msec obtained from 3 electrocardiograms (ECGs); any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec; any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
9. Patients unable to swallow oral medication or patients with GI disorders or significant GI resection likely to interfere with the absorption of AZD9291.
10. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
11. Women who are breastfeeding.
12. Patients with a known hypersensitivity to AZD9291 or rifampicin or any of the excipients of the products.
13. Concomitant medication contraindicated for use with rifampicin (including, but not limited to): cisapride, oral midazolam, nisoldipine, pimozide, quinidine, dofetilide, triazolam, levacetylmethadol (levomethadyl), 3-hydroxy-3-methyl-glutaryl coenzyme A (HMG-CoA)-reductase inhibitors metabolised by CYP3A4, such as lovastatin and simvastatin, ergot alkaloids metabolised by CYP3A4, such as dihydroergotamine, ergometrine (ergonovine), ergotamine and methylergometrine (methylergonovine).
14. For optional genetic research: .Previous allogenic bone marrow transplant or Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, MSD, Study Director — AstraZeneca
Locations (14):
- United States (2):
  - Research Site, Atlanta, Georgia
  - Research Site, Detroit, Michigan
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Research Site, Taipei, Taiwan
- United Kingdom (2):
  - Research Site, Cardiff
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Vishwanathan K, Dickinson PA, So K, Thomas K, Chen YM, De Castro Carpeno J, Dingemans AC, Kim HR, Kim JH, Krebs MG, Chih-Hsin Yang J, Bui K, Weilert D, Harvey RD. The effect of itraconazole and rifampicin on the pharmacokinetics of osimertinib. Br J Clin Pharmacol. 2018 Jun;84(6):1156-1169. doi: 10.1111/bcp.13534. Epub 2018 Mar 23. PMID 29381826
- See also: StudyD5160C00013_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2990&filename=StudyD5160C00013_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 04 December 2014; Last Subject Last Visit Part A: 09 July 2015 and Part B: 29 June 2016. Study performed at 18 sites across Asia, North America and Western Europe. Part A assessed effect of multiple doses of rifampicin on PK of AZD9291; Part B allowed subjects further access to AZD9291 and provided additional safety data.
Pre-assignment Details: 51 patients were enrolled (signed informed consent). Patients were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 10 subjects were enrolled but failed inclusion/exclusion criteria and so were not eligible to be assigned treatment. The remaining 41 patients started Period 1 and received treatment.
Groups:
- AZD9291 and Rifampicin (Part A); AZD9291 Alone (Part B): In Part A of the study, sequential treatments of AZD9291 alone, followed by AZD9291 + rifampicin, followed by AZD9291 alone. Each patient received 80 mg oral doses of AZD9291 tablets once daily for 77 days (Days 1 to 77) and additionally received 600 mg oral doses of rifampicin once daily on Days 29 to 49.
  In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Period: Part A: Day 1-28 (AZD9291 Alone)
Arm/Group | AZD9291 and Rifampicin (Part A); AZD9291 Alone (Part B)
Started | 41
Completed | 41
Not Completed | 0
Period: Part A: Day 29-49 (AZD9291+Rifampicin)
Arm/Group | AZD9291 and Rifampicin (Part A); AZD9291 Alone (Part B)
Started | 41
Completed | 37
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Condition under investigation worsened | 2
Period: Part A: Day 50-77 (AZD9291 Alone)
Arm/Group | AZD9291 and Rifampicin (Part A); AZD9291 Alone (Part B)
Started | 37
Completed | 32
Not Completed | 5
Not completed — Condition under investigation worsened | 5
Period: Part B: Day 78 to End Part B (AZD9291)
Arm/Group | AZD9291 and Rifampicin (Part A); AZD9291 Alone (Part B)
Started | 34 (32 completed Part A + 2 entered Part B without completing Part A (both due to AE) =34 started Part B)
Completed | 19
Not Completed | 15
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Newly discovered brain metastases | 1
Not completed — Death | 1
Not completed — Condition under investigation worsened | 9

BASELINE CHARACTERISTICS:
Population: All patients in the safety analysis set who received at least one dose of AZD9291 (n = 41) were included in the baseline analysis.
Arm/Group | AZD9291 and Rifampicin (Part A); AZD9291 Alone (Part B)
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Maximum Plasma Concentration for AZD9291 After Dosing Alone and in Combination With Rifampicin (Css,Max)
Description: Rate and extent of absorption of AZD9291 by assessment of maximum plasma concentration at steady state (Css,max). AZD9291 doses were first without, then with rifampicin (Periods 1 and 2, respectively).
Time Frame: Samples collected on Day 28 following AZD9291 alone and Day 49 (following AZD9291 and rifampicin) at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose in Part A.
Population: The PK analysis set included all dosed patients who had at least 1 quantifiable plasma concentration collected post-dose without any important deviations or events that would exclude the patient.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Groups:
- AZD9291 Alone (Period 1): AZD9291 80 mg once daily on Days 1 to 28 (Part A). AZD9291 was administered fasted from at least 2 hours before dosing to at least 2 hours after dosing. Water was allowed as desired except for 1 hour before and after AZD9291 administration on Day 28.
- AZD9291 + Rifampicin (Period 2): Concomitant treatment with AZD9291 80 mg once daily and rifampicin 600 mg once daily on Days 29 to 49 (Part A). All treatments (AZD9291 and rifampicin) were administered fasted from at least 2 hours before dosing to at least 2 hours after dosing. Water was allowed as desired except for 1 hour before and after AZD9291 administration on Day 49.
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 38 | 32
nanomolar (nM) | 577.4 (44.7) | 147.5 (48.2)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 + Rifampicin (Period 2); Natural log-transformed Css,max values were compared between periods using a mixed effects analysis of variance (ANOVA) with period as fixed effect and patient as random effect. It was assumed the within-patient coefficient of variation for AZD9291 in both area under the plasma concentration-time curve during the dosing interval (AUCtau) and Cmax was 34%. A 33% decrease in exposure for AZD9291 when given with rifampicin was also assumed; Test type: Non-Inferiority or Equivalence — No effect on the PK of AZD9291 after co-administration of rifampicin was concluded if the lower bound of the 90% confidence intervals (CIs) for the ratios (Period 2 versus Period 1) of AZD9291 AUCtau and Css,max were both above 50%. The experiment-wide power for the ratios being above 50% was 90% (95% power for each parameter); Geometric least-squares (LS) mean ratio = 27.16, 90% CI 2-sided [24.36 to 30.29] — AZD9291+rifampicin / AZD9291 alone (Period 2 versus Period 1)

2. Primary Outcome: Assessment of Area Under the Plasma Concentration-time Curve During the Dosing Interval for AZD9291 After Dosing Alone and in Combination With Rifampicin (AUCtau)
Description: Rate and extent of absorption of AZD9291 by assessment of AUCtau. AZD9291 doses were first without, then with rifampicin (Periods 1 and 2, respectively).
Time Frame: Samples collected on Day 28 following AZD9291 alone and Day 49 following AZD9291 and rifampicin at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose in Part A.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM * hour (nM*h)
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 38 | 32
nM * hour (nM*h) | 10870 (44.3) | 2192 (43.8)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 + Rifampicin (Period 2); Natural log-transformed AUCtau values were compared between periods using a mixed effects ANOVA with period as fixed effect and patient as random effect. It was assumed the within-patient coefficient of variation for AZD9291 in both AUCtau and Cmax was 34%. A 33% decrease in exposure for AZD9291 when given with rifampicin was also assumed; Test type: Non-Inferiority or Equivalence — No effect on the PK of AZD9291 after co-administration of rifampicin was concluded if the lower bound of the 90% CIs for the ratios (Period 2 versus Period 1) of AZD9291 AUCtau and Css,max were both above 50%. The experiment-wide power for the ratios being above 50% was 90% (95% power for each parameter); Geometric LS Mean Ratio = 21.55, 90% CI 2-sided [19.50 to 23.83] — AZD9291+rifampicin / AZD9291 alone (Period 2 versus Period 1)

3. Secondary Outcome: Assessment of Css,Max for AZD9291 Before and After Rifampicin
Description: Rate and extent of absorption of AZD9291 by assessment of Css,max. AZD9291 alone before rifampicin (Period 1) and AZD9291 alone after rifampicin (Period 3).
Time Frame: Samples collected on Day 28 and 77 following AZD9291 alone at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose in Part A.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- AZD9291 Alone (Period 3): AZD9291 80 mg once daily on Days 50 to 77 (Part A). AZD9291 was administered fasted from at least 2 hours before dosing to at least 2 hours after dosing. Water was allowed as desired except for 1 hour before and after AZD9291 administration on Day 77.
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 28
nM | 577.4 (44.7) | 531.4 (37.9)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 Alone (Period 3); Natural log-transformed Css,max values were compared between periods using a mixed effects ANOVA with period as a fixed effect and patient as a random effect; Test type: Superiority or Other; Geometric LS Mean Ratio = 95.53, 90% CI 2-sided [85.27 to 107.03] — AZD9291 alone / AZD9291 alone (Period 3 versus Period 1). No pre-specified margins for equivalence test for AZD9291 alone in separate periods, but analysed for consistency with AZD9291+rifampicin / AZD9291 alone analysis (primary outcome measure)

4. Secondary Outcome: Assessment of Css,Max for AZ5104 (Metabolite)
Description: Rate and extent of absorption of AZ5104 (metabolite) by assessment of Css,max. AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: Samples collected on Day 28 and 77 (following AZD9291 alone) and Day 49 (following AZD9291 and rifampicin) at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose in Part A.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
nM | 60.40 (57.2) | 12.28 (52.6) | 50.73 (49.8)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 + Rifampicin (Period 2); For AZ5104 (metabolite), natural log-transformed Css,max values were compared between periods using a mixed effects ANOVA with period as a fixed effect and patient as a random effect; Test type: Superiority or Other; Geometric LS Mean Ratio = 21.72, 90% CI 2-sided [19.08 to 24.72] — AZD9291+rifampicin / AZD9291 alone (Period 2 versus Period 1). No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis
Statistical Analysis 2: Comparison: AZD9291 Alone (Period 1) vs AZD9291 Alone (Period 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric LS Mean Ratio = 88.31, 90% CI 2-sided [77.17 to 101.07] — AZD9291 alone / AZD9291 alone (Period 3 versus Period 1). No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis

5. Secondary Outcome: Assessment of Css,Max for AZ7550 (Metabolite)
Description: Rate and extent of absorption of AZ7550 (metabolite) by assessment of Css,max. AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
nM | 53.54 (43.7) | 73.14 (25.0) | 53.24 (34.4)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 + Rifampicin (Period 2); For AZ7550 (metabolite), natural log-transformed Css,max values were compared between periods using a mixed effects ANOVA with period as a fixed effect and patient as a random effect; Test type: Superiority or Other; Geometric LS Mean Ratio = 139.32, 90% CI 2-sided [127.74 to 151.96] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: AZD9291 Alone (Period 1) vs AZD9291 Alone (Period 3); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Geometric LS Mean Ratio = 100.75, 90% CI 2-sided [92.04 to 110.29] — [estimate comment as in outcome 4, analysis 2]

6. Secondary Outcome: Assessment of Css,Max for Rifampicin
Description: Rate and extent of absorption of rifampicin by assessment of Css,max. AZD9291 dosing in combination with rifampicin (Period 2).
Time Frame: Samples collected on Day 49 (following AZD9291 and rifampicin) at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose in Part A.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 32
nanogram per millilitre (ng/mL) | 13810 (40.6)

7. Secondary Outcome: Assessment of AUCtau for AZD9291 Before and After Rifampicin
Description: Rate and extent of absorption of AZD9291 by assessment of AUCtau. AZD9291 alone before rifampicin (Period 1) and AZD9291 alone after rifampicin (Period 3).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 28
nM*h | 10870 (44.3) | 10060 (36.8)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 Alone (Period 3); Natural log-transformed AUCtau values were compared between periods using a mixed effects ANOVA with period as a fixed effect and patient as a random effect; Test type: Superiority or Other; Geometric LS Mean Ratio = 95.89, 90% CI 2-sided [86.37 to 106.45] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Assessment of AUCtau for AZ5104 (Metabolite)
Description: Rate and extent of absorption of AZ5104 (metabolite) by assessment of AUCtau. AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
nM*h | 1206 (55.8) | 210.3 (48.0) | 1029 (49.7)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 + Rifampicin (Period 2); For AZ5104 (metabolite), natural log-transformed AUCtau values were compared between periods using a mixed effects ANOVA with period as a fixed effect and patient as a random effect; Test type: Superiority or Other; Geometric LS Mean Ratio = 18.76, 90% CI 2-sided [16.61 to 21.19] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: AZD9291 Alone (Period 1) vs AZD9291 Alone (Period 3); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; Geometric LS Mean Ratio = 90.08, 90% CI 2-sided [79.34 to 102.27] — [estimate comment as in outcome 4, analysis 2]

9. Secondary Outcome: Assessment of AUCtau for AZ7550 (Metabolite)
Description: Rate and extent of absorption of AZ7550 (metabolite) by assessment of AUCtau. AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
nM*h | 1107 (41.7) | 1416 (25.6) | 1111 (31.7)
Statistical Analysis 1: Comparison: AZD9291 Alone (Period 1) vs AZD9291 + Rifampicin (Period 2); For AZ7550 (metabolite), natural log-transformed AUCtau values were compared between periods using a mixed effects ANOVA with period as a fixed effect and patient as a random effect; Test type: Superiority or Other; Geometric LS Mean Ratio = 129.81, 90% CI 2-sided [119.14 to 141.44] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: AZD9291 Alone (Period 1) vs AZD9291 Alone (Period 3); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Geometric LS Mean Ratio = 100.76, 90% CI 2-sided [92.15 to 110.19] — [estimate comment as in outcome 4, analysis 2]

10. Secondary Outcome: Assessment of AUCtau for Rifampicin
Description: Rate and extent of absorption of rifampicin by assessment of AUCtau. AZD9291 dosing in combination with rifampicin (Period 2).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 32
ng*h/mL | 58610 (36.8)

11. Secondary Outcome: Assessment of Tss,Max for AZD9291, and AZ5104 and AZ7550 (Metabolites)
Description: Rate and extent of absorption of AZD9291, and AZ5104 and AZ7550 (metabolites) by assessment of time to reach maximum plasma concentration at steady state (tss,max). AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
h
  AZD9291 tss,max | 4.97 [2.88 to 9.88] | 5.88 [3.00 to 10.00] | 6.00 [3.17 to 23.92]
  AZ5104 tss,max | 6.00 [0.00 to 24.00] | 6.03 [3.00 to 11.43] | 6.00 [0.00 to 24.00]
  AZ7550 tss,max | 6.14 [2.88 to 24.92] | 7.95 [4.00 to 12.00] | 7.03 [1.10 to 24.00]

12. Secondary Outcome: Assessment of Tss,Max for Rifampicin
Description: Rate and extent of absorption of rifampicin by assessment of tss,max. AZD9291 dosing in combination with rifampicin (Period 2).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 32
h | 2.00 [0.83 to 6.07]

13. Secondary Outcome: Assessment of Css,Min for AZD9291, and AZ5104 and AZ7550 (Metabolites)
Description: Rate and extent of absorption of AZD9291, and AZ5104 and AZ7550 (metabolites) by assessment of minimum plasma concentration at steady state (Css,min). AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 31 | 28
nM
  AZD9291 Css,min | 354.7 (52.4) | 50.56 (47.9) | 326.9 (41.1)
  AZ5104 Css,min | 41.80 (62.1) | 5.816 (51.6) | 35.37 (51.4)
  AZ7550 Css,min | 37.99 (44.0) | 44.89 (26.9) | 37.68 (35.4)

14. Secondary Outcome: Assessment of Css,Min for Rifampicin
Description: Rate and extent of absorption of rifampicin by assessment of minimum plasma concentration at steady state (Css,min). AZD9291 dosing in combination with rifampicin (Period 2).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 32
ng/mL | NA (NA) — Geometric mean and percent geometric coefficient of variation were not determined for Css,min for rifampicin since a number of patients had concentration values below the limits of quantitation at the end of the 24 hour dosing interval.

15. Secondary Outcome: Assessment of CLss/F for AZD9291
Description: Rate and extent of absorption of AZD9291 by assessment of the apparent plasma clearance following oral administration and multiple dosing (CLss/F). AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre per hour (L/h)
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
Litre per hour (L/h) | 14.74 (44.2) | 73.07 (43.8) | 15.92 (36.7)

16. Secondary Outcome: Assessment of CLss/F for Rifampicin
Description: Rate and extent of absorption of rifampicin by assessment of CLss/F. AZD9291 dosing in combination with rifampicin (Period 2).
Time Frame: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | AZD9291 + Rifampicin (Period 2)
Number analyzed (Participants) | 32
L/h | 10.23 (36.7)

17. Secondary Outcome: Assessment of the Metabolic Ratios of Css,Max for AZ5104 and AZ7550 (MRCss,Max)
Description: Assessment of the metabolite to parent ratio (calculated as AZ5104 to AZD9291 and AZ7550 to AZD9291) for Css,max (MRCss,max). AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
Ratio
  AZ5104 Css,max / AZD9291 Css,max | 0.1046 (31.0) | 0.08327 (27.4) | 0.09544 (27.4)
  AZ7550 Css,max / AZD9291 Css,max | 0.09276 (49.3) | 0.4960 (33.1) | 0.1002 (38.1)

18. Secondary Outcome: Assessment of the Metabolic Ratios of AUCtau for AZ5104 and AZ7550 (MRAUCtau)
Description: Assessment of the metabolite to parent ratio (calculated as AZ5104 to AZD9291 and AZ7550 to AZD9291) for AUCtau (MRAUCtau). AZD9291 dosing alone and in combination with rifampicin (all periods).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD9291 Alone (Period 1) | AZD9291 + Rifampicin (Period 2) | AZD9291 Alone (Period 3)
Number analyzed (Participants) | 38 | 32 | 28
Ratio
  AZ5104 AUCtau / AZD9291 AUCtau | 0.1109 (29.0) | 0.09595 (23.6) | 0.1023 (28.5)
  AZ7550 AUCtau / AZD9291 AUCtau | 0.1019 (52.3) | 0.6459 (28.2) | 0.1104 (38.8)

ADVERSE EVENTS:
Time Frame: Approximately 3 months for Part A; up to approximately 14 months for Part B and approximately 17 months for Overall (Parts A and B combined).
Description: Part A: Adverse events (AEs) collected from day of first dose until day prior to first dose in Part B (Day 77), or until 30 days after last dose if discontinued in Part A.
  Part B: AEs collected from day of first dose in Part B until 30 days after last dose, or until last dose in Part B for those entering continued access phase (CAP).
Groups:
- Overall: Parts A and B of the study combined.
- Part A: In Part A of the study, each patient received 80 mg oral doses of AZD9291 tablets once daily for 77 days (Days 1 to 77) and additionally received 600 mg oral doses of rifampicin once daily on Days 29 to 49.
- Part B: In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Arm/Group | Overall | Part A | Part B
Serious Adverse Events (participants affected / at risk) | 11/41 | 7/41 | 6/34
Other Adverse Events (participants affected / at risk) | 40/41 | 39/41 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=41) | Part A (N=41) | Part B (N=34)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=41) | Part A (N=41) | Part B (N=34)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 3 (3)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (10) | 4 (4) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 22 (39) | 14 (18) | 14 (21)
Oedema peripheral (General disorders) | 7 (7) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4) | 2 (2)
Weight decreased (Investigations) | 7 (7) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 19 (22) | 6 (8) | 13 (14)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 2 (2) | 2 (3)
Dry eye (Eye disorders) | 4 (5) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 2 (2) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (24) | 8 (14) | 9 (10)
Stomatitis (Gastrointestinal disorders) | 10 (14) | 6 (6) | 6 (8)
Vomiting (Gastrointestinal disorders) | 11 (16) | 5 (7) | 7 (9)
Asthenia (General disorders) | 7 (8) | 4 (5) | 3 (3)
Face oedema (General disorders) | 3 (3) | 2 (2) | 1 (1)
Fatigue (General disorders) | 13 (14) | 8 (9) | 5 (5)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 5 (6) | 1 (1) | 4 (5)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Paronychia (Infections and infestations) | 8 (13) | 2 (2) | 6 (11)
Urinary tract infection (Infections and infestations) | 6 (12) | 6 (6) | 2 (6)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 2 (3)
Blood creatinine increased (Investigations) | 3 (4) | 1 (1) | 2 (3)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 3 (6) | 2 (3) | 2 (3)
Platelet count decreased (Investigations) | 5 (7) | 2 (3) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (17) | 6 (8) | 5 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (6) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 8 (13) | 7 (10) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 7 (7) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 3 (4) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (27) | 10 (12) | 12 (15)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (4) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 4 (7) | 4 (4) | 1 (3)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
At end of Part B, the CAP allowed patients to continue receiving AZD9291 if still deriving clinical benefit. No clinical data was databased during the CAP; thus AE data is presented to end of Part B only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.